CLINICAL TRIAL: NCT04236245
Title: EU Post Market Clinical Follow-Up Study of the Venclose System for Saphenous Vein Incompetence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venclose, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VENC17A
Record Dates: First submitted 2020-01-14; First posted 2020-01-22 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Chronic Venous Insufficiency
Keywords: GSV; superficial vein reflux; venous reflux; venous insufficiency; varicose veins
MeSH Terms: conditions — Venous Insufficiency; Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Venclose RF System (Other): Treatment of great saphenous vein (GSV) using Venclose RF System
  Interventions: Device: Venclose RF System

INTERVENTIONS:
Device: Venclose RF System — Treatment of great saphenous vein (GSV) using Venclose RF System
  Other Names: RF ablation, EVSRF

SUMMARY:
This is a prospective, non-randomized study in which patients who meet eligibility criteria and consent to participate will undergo a minimally invasive procedure using radiofrequency (RF) energy for ablation of the great saphenous vein (GSV).

DETAILED DESCRIPTION:
Subjects who meet eligibility criteria will undergo a procedure using the Venclose Radiofrequency (RF) System to treat the great saphenous vein.

The technique involves percutaneous access and insertion of the endovenous sectional radiofrequency (EVSRF™) catheter into the target vein under ultrasound guidance and relies on the use of local anesthesia and thermal energy, from a radiofrequency generator, applied to the target vein. After each treatment, the EVSRF™ catheter is withdrawn a single length of the heating coil and another treatment is performed, until the entire vessel has been treated.

After the treatment procedure, subjects will be evaluated four (4) times to assess vein recanalization and reflux, and to determine the incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and 18 to 80 years old (inclusive) at time of enrollment (signing of consent).
* Subject has significant venous reflux by Duplex Ultrasound (DUS), defined as reverse flow with reflux duration greater than 0.5 seconds after the Valsalva maneuver or distal augmentation while the patient is standing or in reverse Trendelenburg position.
* Subject is eligible for endovascular treatment, as determined by the treating investigator.
* Subject's general physical condition allows for a significant amount of ambulation after the procedure, as determined by the treating investigator.
* Subject is willing and able to complete study requirements, including all follow-up visits and assessments.
* Subject voluntarily provides written informed consent to participate in this study.

Exclusion Criteria:

* There is evidence of old or fresh thrombus in the subject's diseased vein segment to be treated, as determined by Duplex Ultrasound (DUS) within 2 weeks prior to the index procedure.
* In the judgment of the treating investigator heat energy delivery to the subject would be contraindicated.
* Subject is concurrently participating in another interventional clinical trial.
* Subject is pregnant or plans to be pregnant or lactating at the time of the treatment procedure.
* Subject has known or suspected allergies or contraindications to any general or local anesthetic agents and/or any antibiotic medication that cannot be adequately pre-treated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mattausch, Dr. med, Principal Investigator — Venenzentrum am Bruehl
Locations (1):
- Venenzentrum am Bruehl, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasquez MA, Rabe E, McLafferty RB, Shortell CK, Marston WA, Gillespie D, Meissner MH, Rutherford RB; American Venous Forum Ad Hoc Outcomes Working Group. Revision of the venous clinical severity score: venous outcomes consensus statement: special communication of the American Venous Forum Ad Hoc Outcomes Working Group. J Vasc Surg. 2010 Nov;52(5):1387-96. doi: 10.1016/j.jvs.2010.06.161. Epub 2010 Sep 27. PMID 20875713

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Venclose RF System
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 25

OUTCOME MEASURES:

1. Primary Outcome: Vein Occlusion Rate
Description: Percentage of limbs with occlusion of the treated vein
Time Frame: 3 days
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (limbs) | 29
limbs
  Complete Occlusion | 29
  Segmental Recanalization | 0
  Complete Recanalization | 0

2. Primary Outcome: Vein Occlusion Rate
Description: Percentage of limbs with occlusion of the treated vein
Time Frame: 3 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  Complete Occlusion | 28
  Segmental Recanalization | 1
  Complete Recanalization | 0

3. Primary Outcome: Vein Occlusion Rate
Description: Percentage of limbs with occlusion of the treated vein
Time Frame: 6 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  Complete Occlusion | 28
  Segmental Recanalization | 1
  Complete Recanalization | 0

4. Primary Outcome: Vein Occlusion Rate
Description: Percentage of limbs with occlusion of the treated vein
Time Frame: 12 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  Complete Occlusion | 28
  Segmental Recanalization | 1
  Complete Recanalization | 0

5. Primary Outcome: Reflux-free Rate
Description: Percentage of limbs without reflux in the treated vein
Time Frame: 3 days
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  No reflux along treated GSV | 29
  Reflux along treated GSV | 0

6. Primary Outcome: Reflux-free Rate
Description: Percentage of limbs without reflux in the treated vein
Time Frame: 3 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  No reflux along treated GSV | 28
  Reflux along treated GSV | 1

7. Primary Outcome: Reflux-free Rate
Description: Percentage of limbs without reflux in the treated vein
Time Frame: 6 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  No reflux along treated GSV | 28
  Reflux along treated GSV | 1

8. Primary Outcome: Reflux-free Rate
Description: Percentage of limbs without reflux in the treated vein
Time Frame: 12 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  No reflux along treated GSV | 28
  Reflux along treated GSV | 1

9. Secondary Outcome: Clinical Etiologic Anatomic Pathophysiologic (CEAP) Classification
Description: Clinical signs and symptoms of lower limb venous disease (Scale C0-C6: MIN: C0=no visible or palpable signs of venous disease; MAX: C6=active venous ulcer)
Time Frame: Baseline
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  C0: No visible or palpable signs of venous disease | 0
  C1: Telangiectasies or reticular veins | 0
  C2: Varicose veins | 0
  C3: Edema | 24
  C4a: Pigmentation or eczema | 4
  C4b: Lipodermatosclerosis or atrophie blanche | 0
  C5: Healed venous ulcer | 1
  C6: Active venous ulcer | 0

10. Secondary Outcome: Clinical Etiologic Anatomic Pathophysiologic (CEAP) Classification
Description: as for outcome 9
Time Frame: 3 days
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  C0: No visible or palpable signs of venous disease | 0
  C1: Telangiectasies or reticular veins | 1
  C2: Varicose veins | 0
  C3: Edema | 24
  C4a: Pigmentation or eczema | 3
  C4b: Lipdermatosclerosis or atrophie blanche | 0
  C5: Healed venous ulcer | 1
  C6: Active venous ulcer | 0

11. Secondary Outcome: Clinical Etiologic Anatomic Pathophysiologic (CEAP) Classification
Description: Clinical signs and symptoms of lower limb venous disease (Scale C0-C6: MIN: C0=no visible or palpable signs of venous disease; MAX: C6=active venous ulcer
Time Frame: 3 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  C0: No visible or palpable signs of venous disease | 1
  C1: Telangiectasies or reticular veins | 11
  C2: Varicose veins | 10
  C3: Edema | 4
  C4a: Pigmentation or eczema | 2
  C4b: Lipodermatosclerosis or atrophie blanche | 0
  C5: Healed venous ulcer | 1
  C6: Active venous ulcer | 0

12. Secondary Outcome: Clinical Etiologic Anatomic Pathophysiologic (CEAP) Classification
Description: as for outcome 9
Time Frame: 6 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  C0: No visible or palpable signs of venous disease | 1
  C1: Telangiectasies or reticular veins | 19
  C2: Varicose veins | 5
  C3: Edema | 1
  C4a: Pigmentation or eczema | 2
  C4b: Lipodermatosclerosis or atrophie blanche | 0
  C5: Healed venous ulcer | 1
  C6: Active venous ulcer | 0

13. Secondary Outcome: Clinical Etiologic Anatomic Pathophysiologic (CEAP) Classification
Description: as for outcome 9
Time Frame: 12 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  C0: No visible or palpable signs of venous disease | 1
  C1: Telangiectasies or reticular veins | 21
  C2: Varicose veins | 3
  C3: Edema | 1
  C4a: Pigmentation or eczema | 2
  C4b: Lipodermatosclerosis or atrophie blanche | 0
  C5: Healed venous ulcer | 1
  C6: Active venous ulcer | 0

14. Secondary Outcome: Venous Clinical Severity Score (VCSS)
Description: Assessment of venous disease (Scale 0-30: MIN=0 (least severe); MAX=30 (most severe))
Time Frame: Baseline
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
score on a scale | 4.4 (1.8)

15. Secondary Outcome: Venous Clinical Severity Score (VCSS)
Description: Assessment of venous disease (Scale 0-30: MIN=0 (least severe); MAX=30 (most severe))
Time Frame: 3 days
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
score on a scale | 5.9 (1.1)

16. Secondary Outcome: Venous Clinical Severity Score (VCSS)
Description: Assessment of venous disease (Scale 0-30: MIN=0 (least severe); MAX=30 (most severe))
Time Frame: 3 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
score on a scale | 1.6 (1.3)

17. Secondary Outcome: Venous Clinical Severity Score (VCSS)
Description: Assessment of venous disease (Scale 0-30: MIN=0 (least severe); MAX=30 (most severe))
Time Frame: 6 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
score on a scale | 0.7 (1.0)

18. Secondary Outcome: Venous Clinical Severity Score (VCSS)
Description: Assessment of venous disease (Scale 0-30: MIN=0 (least severe); MAX=30 (most severe))
Time Frame: 12 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
score on a scale | 0.6 (0.9)

19. Secondary Outcome: Presence of Complications From GSV Intervention
Description: Number of limbs that presented with the listed complications and side effects resulting from the GSV intervention
Time Frame: up to 3 days
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Number; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  Allergic reaction to local anesthesia | 0
  Allergic reaction to device | 0
  Vein perforation | 0
  Thermal skin injury | 0
  Skin discoloration or pigmentation | 0
  Infection | 0
  Neurological injury | 0
  Paresthesia | 1
  Superficial venous thrombophlebitis | 0
  Edema | 0
  Ecchymosis | 0
  Hematoma | 0
  Erythema | 0
  EHIT II (non-occlusive DVT) | 1
  Deep vein thrombosis (DVT) or pulmonary embolism (PE) | 0

20. Secondary Outcome: Presence of Complications From GSV Intervention
Description: Number of limbs that presented with the listed complications and side effects resulting from the GSV intervention
Time Frame: 3 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Number; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  Allergic reaction to local anesthesia | 0
  Allergic reaction to device | 0
  Vein perforation | 0
  Thermal skin injury | 0
  Skin discoloration or pigmentation | 0
  Infection | 0
  Neurological injury | 0
  Paresthesia | 0
  Superficial venous thrombophlebitis | 0
  Edema | 0
  Ecchymosis | 0
  Hematoma | 0
  Erythema | 0
  EHIT II (non-occlusive DVT) | 0
  Deep vein thrombosis (DVT) or pulmonary embolism (PE) | 0

21. Secondary Outcome: Presence of Complications From GSV Intervention
Description: Number of limbs that presented with the listed complications and side effects resulting from the GSV intervention
Time Frame: 6 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Number; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  Allergic reaction to local anesthesia | 0
  Allergic reaction to device | 0
  Vein perforation | 0
  Thermal skin injury | 0
  Skin discoloration or pigmentation | 0
  Infection | 0
  Neurological injury | 0
  Paresthesia | 0
  Superficial venous thrombophlebitis | 0
  Edema | 0
  Ecchymosis | 0
  Hematoma | 0
  Erythema | 0
  EHIT II (non-occlusive DVT) | 0
  Deep vein thrombosis (DVT) or pulmonary embolism (PE) | 0

22. Secondary Outcome: Presence of Complications From GSV Intervention
Description: Number of limbs that presented with the listed complications and side effects resulting from the GSV intervention
Time Frame: 12 months
Population: Twenty-five subjects were treated, 4 of whom were treated bilaterally, for a total of 29 limbs treated.
Measure: Number; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Venclose RF System
Number analyzed (Participants) | 25
Number analyzed (Limbs) | 29
Limbs
  Allergic reaction to local anesthesia | 0
  Allergic reaction to device | 0
  Vein perforation | 0
  Thermal skin injury | 0
  Skin discoloration or pigmentation | 0
  Infection | 0
  Neurological injury | 0
  Paresthesia | 0
  Superficial venous thrombophlebitis | 0
  Edema | 0
  Ecchymosis | 0
  Hematoma | 0
  Erythema | 0
  EHIT II (non-occlusive DVT) | 0
  Deep vein thrombosis (DVT) or pulmonary embolism (PE) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from time of treatment through one year.
Arm/Group | Venclose RF System
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 5/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venclose RF System (N=25)
Non-occlusive DVT (Vascular disorders) | 2 (2)
Muscle vein thrombosis (Vascular disorders) | 1 (1)
Pain (Vascular disorders) | 1 (1)
Lymphedema (Blood and lymphatic system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT04236245/Prot_SAP_000.pdf